CLINICAL TRIAL: NCT00636844
Title: Detection of Chemotherapy Induced Cardiotoxicity
Status: Completed | Type: Observational
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Other Study IDs: JL-001
Record Dates: First submitted 2008-03-10; First posted 2008-03-17 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2012-08

CONDITIONS: Cancer
Keywords: chemotherapy, cardiotoxicity
MeSH Terms: conditions — Neoplasms; Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample for analysis of mRNA and oxidative stress markers
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group A: Patients receiving chemotherapy (anthracycline and/or adjuvant trastuzumab) for the first time

SUMMARY:
To identify patients that are at risk of heart damage after receiving chemotherapy (adriamycin).

DETAILED DESCRIPTION:
To identify patients at risk of development of heart damage after receiving chemotherapy by obtaining the genetic profile of those who show: elevation of troponin, left ventricular systolic and diastolic dysfunction, and pro-oxidant stress markers.

ELIGIBILITY:
Inclusion Criteria:

* undergoing anthracycline and/or trastuzumab therapy for the first time

Exclusion Criteria:

* abnormal ventricular ejection fraction
* past history of, or active cardiac disease including: MI, CHF, angina, arrhythmia requiring medication, valvular disease, uncontrolled systemic hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oncology clinic patients
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The genetic profile of patients with anthracycline-induced elevation of troponin-I | one year

SECONDARY OUTCOMES:
Assess the genetic profile of patient with anthracycline-induced left ventricular systolic and diastolic dysfunction | one year
Assess the relationship of quantitative increases of pro-oxidant stress and a specific genetic profile | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jannet Lewis, MD, Principal Investigator — George Washington University
Locations (1):
- George Washington University, Washington D.C., District of Columbia, United States